CLINICAL TRIAL: NCT03481101
Title: WHENII - Early Response Evaluation With 18F-2-fluoro-2-deoxy-D-glucose Fluorodeoxyglucose(FDG)- Positrons Emissions Tomography(PET)/CT and Liquid Biopsy in Patients With NSCLC (Non Small Cell Lung Cancer)
Brief Title: WHENII - Early Response Evaluation With FDG-PET/CT and Liquid Biopsy in Patients With NSCLC
Acronym: WHENII
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, heidi ryssel, Doctor, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H-17016437
Record Dates: First submitted 2018-03-05; First posted 2018-03-29 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Non Small Cell Lung Cancer; Circulating Tumor Cell; Circulating Tumor DNA
Keywords: early response evaluation; immunotherapy; chemotherapy; liquid biopsy; FDG-PET/CT
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplastic Cells, Circulating | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Intervention Model Description: response evaluation with FDG-PET and free circulating DNA in patients with inoperable lung cancer of non small cell type during first treatment with chemotherapy or immunotherapy.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All patients (Other): Both patients receiving chemotherapy and immunotherapy are observed during the same intervention with PET/CT and liquid biopsy. No primary comparison are made between the groups.
  Interventions: Device: PET/CT

INTERVENTIONS:
Device: PET/CT — 3 extra scans with FDG-PET/CT and 4 blood samples

SUMMARY:
Response evaluation with FDG-PET and free circulating DNA in patients with inoperable lung cancer of non small cell type during first treatment with chemotherapy or immunotherapy.

DETAILED DESCRIPTION:
Interventional study of patients with inoperable lung cancer of non small cell type undergoing 1st treatment of either chemotherapy or immunotherapy. Patients are evaluated with FDG-PET/ct and blood analyses og circulating tumor DNA and cancer markers to determine early response.

PET-CT are preceded before and after treatment is given;

* day 0 before treatment,
* day 2 after treatment and
* day 21 just before second treatment. At every FDG-PET/ct scan blood are examined for circulating tumor DNA (ctDNA) and potentially cancer markers by White genome sequencing. In total 3 PET-CT scans and 4 blood samples are performed. The result are compared with the standard CT scan after 2-3 cycles of treatment. Blood analyses are repeated after 2-3 cycles to observe any changes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-small cell lung cancer (NSCLC) who is about to start treatment with chemo- or immune therapy. No prior treatment of the one given.
* Measurable decease according to RECIST criteria
* Age > 18 years
* Performance status 0-2 (0-1 for immunotherapy)
* Understands and reads danish

Exclusion Criteria:

* Poor performance status
* Secondary active cancer
* Pregnancy
* Dysregulated diabetes mellitus

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-02-28 (Actual); Primary Completion 2021-02-26 (Estimated); Study Completion 2021-02-28 (Estimated)

PRIMARY OUTCOMES:
Observation of changes in metabolism in cancer cells during first treatment with chemotherapy or immunotherapy. | 3 months
  Measure changes in standardized uptake value (SUV) in tumorcells by FDG-PET.
Observation of changes in circulating tumor DNA during first treatment. | 3 months
  Measure changes in the amount of free circulating DNA
Observation of changes in circulating tumor DNA during first treatment. | 3 months
  Measure changes in cancer DNA by whole genome sequencing on free circulating DNA.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Kjær, Study Director — Klinisk fysiologisk og Nuclearmedicinsk afd
Locations (2):
- Denmark (2):
  - University Copenhagen, Copenhagen
  - University of Copenhagen, Copenhagen

IPD SHARING:
Plan to Share IPD: Undecided